CLINICAL TRIAL: NCT04612608
Title: Assessing the Role of Inclined Positioning in Acute Respiratory Distress Syndrome Patients Recovery
Acronym: ARISE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peter Morris (Other)
Responsible Party: Sponsor-Investigator, Peter Morris, Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 60328
Record Dates: First submitted 2020-10-06; First posted 2020-11-03 (Actual); Last update posted 2022-04-12 (Actual); Status verified 2022-04

CONDITIONS: ARDS, Human
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Intervention Model Description: The intervention arm will undergo a protocol of 4x per day bed elevation to 60 degrees for 30 minutes.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Usual Care
- Intervention (Active Comparator): Intervention arm
  Interventions: Procedure: upright bed

INTERVENTIONS:
Procedure: upright bed — moving the bed into an upright position
  Arms: Intervention

SUMMARY:
The purpose of this study is to determine the effect of intermittent, nearly vertical, patient positioning in a specialized upright bed, on outcomes of mechanically ventilated patients with acute respiratory distress syndrome (ARDS) who are in the ICU.

DETAILED DESCRIPTION:
The purpose of this study is to determine the effect of intermittent, nearly vertical, patient positioning in a specialized upright bed, on outcomes of mechanically ventilated patients with acute respiratory distress syndrome (ARDS) who are in the ICU. This study is a prospective, non-blinded, feasibility, randomized study of ARDS patients, who will be randomized into two treatment groups. One treatment arm will deliver scheduled sessions of upright bed positioning (study intervention), while the other treatment arm receives routine bed position care (care provided exclusively with the bed in the supine position). ICU Practitioners know that positional changes improve clinical outcomes when turning patients from supine to prone (back to belly); however, other positional changes including upright positioning are far less studied. It is well known that in ARDS patients who become proned, an improvement in aeration occurs in the dorsal lung regions (prone positioning has been shown to reduce ARDS mortality). Thus the investigators predict that in this study, the upright positioning holds the potential to further recruit collapsed lung areas. Augmentation of aerated lung while in the upright position is expected to increase the highest value measured per ventilator day of the respiratory system compliance in the upright bed position arm, in a greater fashion than the highest value measured per ventilator day of daily total respiratory system compliance for the usual care arm.

ELIGIBILITY:
Inclusion Criteria:

* Berlin criteria ARDS

Exclusion Criteria:

* ARDS greater than 72 hours
* Neurologic disease known to prolong weaning
* Pregnancy
* Known diagnosis of pulmonary fibrosis
* Implanted cardiac pacer/defibrillator
* prisoner

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2021-05-26 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-01-01 (Actual)

PRIMARY OUTCOMES:
highest value per day of mechanical ventilation of total respiratory system compliance | from the day of randomization, every day of mechanical ventilation until death or liberation from mechanical ventilation up to day 28
  total respiratory system compliance measured 4x daily for each day of mechanical ventilation

CONTACTS AND LOCATIONS:
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: Yes
Investigators will plan to make individual participant data (IPD) available to other researchers
Supporting Information: Study Protocol, SAP, CSR
Time Frame: The data will be available one year following initial study publication for an additional one year
Access Criteria: Discussion of purpose of request with the primary investigator